CLINICAL TRIAL: NCT00372255
Title: An Open, Phase IV Study on the Immunogenicity and Tolerability of Influsplit SSW® 2005/2006 in Children Aged 6 - 13 Years
Brief Title: Study on the Immunogenicity and Tolerability of Influsplit SSW® 2005/2006 in Children Aged 6 - 13 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106252; 2005-004517-14 (EudraCT Number)
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Influsplit SSW® 2005/2006 6-9 years Group (Experimental): Subjects aged 6 to 9 years who received 2 doses of Influsplit SSW® 2005/2006 vaccine at an interval of 4 weeks (Day 0 and Day 28 ± 2).
  Interventions: Biological: Influsplit SSW® 2005/2006
- Influsplit SSW® 2005/2006 10-13 years Group (Active Comparator): Subjects aged 10 to 13 years who received 1 dose of Influsplit SSW® 2005/2006 vaccine at Day 0.
  Interventions: Biological: Influsplit SSW® 2005/2006

INTERVENTIONS:
Biological: Influsplit SSW® 2005/2006 — Study influenza vaccine was administered intramuscularly in the non-dominant arm

SUMMARY:
The study will evaluate the immune response and the tolerability of the influenza vaccine administered in children aged 6-13 years old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children or children with an increased health risk due to an underlying chronic disease-such as chronic airways diseases (including asthma), chronic cardiovascular, hepatic and renal diseases as well as diabetes and other metabolic diseases-aged between 6 and 13 years.
* All subjects must not have received a prior influenza vaccination.
* All subjects must not have had a prior influenza disease.

Exclusion Criteria:

* Use of any study or unlicensed medications/ vaccine other than the study vaccine within 30 days of the vaccination and/or during the study period.
* Acute illness at the start of the study.
* Acute, clinically significant pulmonary, cardiovascular abnormalities or abnormalities of the hepatic or renal function.
* Known allergic reactions which might be caused by the ingredients of the vaccine.
* Girls post-menarche: pregnancy or positive pregnancy-test
* Multiple sclerosis or congenital or acquired immunodeficiencies.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2005-11-17 (Actual); Primary Completion 2006-03-28 (Actual); Study Completion 2006-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Germany (12):
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Bützow, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bischofswerda, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Wurzen, Saxony
  - GSK Investigational Site, Bredstedt, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Niebüll, Schleswig-Holstein
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Schmidt-Ott R, Schwarz T, Haase R, Sander H, Walther U, Fourneau M, Htun-Myint L, Sanger R, Schuster V. Immunogenicity and reactogenicity of a trivalent influenza split vaccine in previously unvaccinated children aged 6-9 and 10-13 years. Vaccine. 2007 Dec 21;26(1):32-40. doi: 10.1016/j.vaccine.2007.10.049. Epub 2007 Nov 9. PMID 18022736
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 106252 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106252 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106252 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106252 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106252 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106252 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by a principal investigator and 22 investigators in 18 centers in Germany.
Groups:
- Influsplit SSW 2005/2006 6-9 Years Group: Subjects aged 6 to 9 years who received 2 doses of Influsplit SSW 2005/2006 vaccine at an interval of 4 weeks (Day 0 and Day 28 ± 2).
- Influsplit SSW 2005/2006 10-13 Years Group: Subjects aged 10 to 13 years who received 1 dose of Influsplit SSW 2005/2006 vaccine at Day 0.
Period: Overall Study
Arm/Group | Influsplit SSW 2005/2006 6-9 Years Group | Influsplit SSW 2005/2006 10-13 Years Group
Started | 110 | 114
Completed | 108 | 113
Not Completed | 2 | 1
Not completed — Withdrawn for other reasons | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influsplit SSW 2005/2006 6-9 Years Group | Influsplit SSW 2005/2006 10-13 Years Group | Total
Number analyzed (Participants) | 110 | 114 | 224
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.4 (1.13) | 11.3 (1.07) | 9.4 (2.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 65 | 127
  Male | 48 | 49 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 107 | 111 | 218
  Not Specified | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease in Children Aged Between 6 and 9 Years
Description: Titers of serum HI antibodies are presented as geometric mean titers (GMTs) against the three influenza strains contained in the trivalent influenza vaccine Influsplit SSW 2005/2006 (GlaxoSmithKline/SSW) after a single versus after two vaccine doses of Influsplit SSW 2005/2006. The three influenza strains assessed were: A/New Caledonia (H1N1), A/New York (H3N2), B/Jiangsu.
Time Frame: 28 days after Dose 1 (Day 28) and 21 days after Dose 2 (Day 49 ± 2)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, included all evaluable subjects for whom data was available for the considered time point and assay assessed.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Influsplit SSW 2005/2006 6-9 Years Group
Number analyzed (Participants) | 97
Titer
  A/New Caledonia (H1N1), Dose 1 | 290.4 [165.6 to 509.3]
  A/New Caledonia (H1N1), Dose 2: number analyzed (Participants) | 95
  A/New Caledonia (H1N1), Dose 2 | 719.2 [503.3 to 1027.7]
  A/New York (H3N2), Dose 1 | 381.2 [281.3 to 516.6]
  A/New York (H3N2), Dose 2: number analyzed (Participants) | 95
  A/New York (H3N2), Dose 2 | 393.9 [313.5 to 494.9]
  B/Jiangsu, Dose 1 | 97.7 [68.6 to 139.2]
  B/Jiangsu, Dose 2: number analyzed (Participants) | 95
  B/Jiangsu, Dose 2 | 301.8 [246.3 to 369.9]

2. Primary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against 3 Strains of Influenza Disease in Children Aged Between 6 and 9 Years
Description: Seroconversion factors were defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The three influenza strains assessed were: A/New Caledonia (H1N1), A/New York (H3N2), B/Jiangsu.
Time Frame: 28 days after Dose 1 (Day 28) and 21 days after Dose 2 (Day 49 ± 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Influsplit SSW 2005/2006 6-9 Years Group
Number analyzed (Participants) | 97
Fold increase
  A/New Caledonia (H1N1), Dose 1 | 16.7 [11.8 to 23.8]
  A/New Caledonia (H1N1), Dose 2: number analyzed (Participants) | 95
  A/New Caledonia (H1N1), Dose 2 | 40.7 [32.6 to 50.8]
  A/New York (H3N2), Dose 1 | 14.9 [10.9 to 20.3]
  A/New York (H3N2), Dose 2: number analyzed (Participants) | 95
  A/New York (H3N2), Dose 2 | 15.4 [11.9 to 20.0]
  B/Jiangsu, Dose 1 | 8.5 [6.7 to 10.7]
  B/Jiangsu, Dose 2: number analyzed (Participants) | 95
  B/Jiangsu, Dose 2 | 26.1 [21.4 to 31.9]

3. Primary Outcome: Number of Seroconverted Subjects Against 3 Strains of Influenza Disease in Children Aged Between 6 and 9 Years
Description: A seroconverted subject was defined as a subject who was either seronegative prior to the vaccination and had a protective post-vaccination titer of greater than or equal to (≥) 1:40 or who was seropositive prior to the vaccination and had at least a 4-fold increase in the titer as the outcome of the vaccination. The three influenza strains assessed were: A/New Caledonia (H1N1), A/New York (H3N2), B/Jiangsu.
Time Frame: 28 days after Dose 1 (Day 28) and 21 days after Dose 2 (Day 49 ± 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influsplit SSW 2005/2006 6-9 Years Group
Number analyzed (Participants) | 97
Participants
  A/New Caledonia (H1N1), Dose 1 | 63
  A/New Caledonia (H1N1), Dose 2: number analyzed (Participants) | 95
  A/New Caledonia (H1N1), Dose 2 | 93
  A/New York (H3N2), Dose 1 | 79
  A/New York (H3N2), Dose 2: number analyzed (Participants) | 95
  A/New York (H3N2), Dose 2 | 80
  B/Jiangsu, Dose 1 | 66
  B/Jiangsu, Dose 2: number analyzed (Participants) | 95
  B/Jiangsu, Dose 2 | 92

4. Secondary Outcome: Titers for Serum HI Antibodies Against 3 Strains of Influenza Disease in Children Aged Between 10 and 13 Years
Description: as for outcome 1
Time Frame: 21 days post-vaccination (Day 21)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Influsplit SSW 2005/2006 10-13 Years Group
Number analyzed (Participants) | 106
Titres
  A/New Caledonia (H1N1), Dose 1 | 1326.6 [856.7 to 2054.3]
  A/New York (H3N2), Dose 1 | 300.6 [241.5 to 374.2]
  B/Jiangsu, Dose 1 | 218.9 [169.1 to 283.5]

5. Secondary Outcome: SCF for HI Antibodies Against 3 Strains of Influenza Disease in Children Aged Between 10 and 13 Years
Description: Seroconversion factors were defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0.The three influenza strains assessed were: A/New Caledonia (H1N1), A/New York (H3N2), B/Jiangsu.
Time Frame: 21 days post-vaccination (Day 21)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Influsplit SSW 2005/2006 10-13 Years Group
Number analyzed (Participants) | 106
Fold increase
  A/New Caledonia (H1N1), Dose 1 | 50.2 [36.2 to 69.8]
  A/New York (H3N2), Dose 1 | 10.3 [8.2 to 12.8]
  B/Jiangsu, Dose 1 | 12.6 [10.4 to 15.3]

6. Secondary Outcome: Number of Seroconverted Subjects Against 3 Strains of Influenza Disease in Children Aged Between 10 and 13 Years
Description: as for outcome 3
Time Frame: 21 days post-vaccination (Day 21)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influsplit SSW 2005/2006 10-13 Years Group
Number analyzed (Participants) | 106
Participants
  A/New Caledonia (H1N1), Dose 1 | 90
  A/New York (H3N2), Dose 1 | 83
  B/Jiangsu, Dose 1 | 90

7. Secondary Outcome: Number of Seroprotected Subjects Who Were Unprotected at Pre-vaccination Against 3 Influenza Strains in Children Aged Between 10 and 13 Years
Description: Seroprotection power (SPP) was defined as the proportion of the subjects unprotected before vaccination (titre < 40) who were protected after vaccination (titer ≥ 40). The three influenza strains assessed were: A/New Caledonia (H1N1), A/New York (H3N2), B/Jiangsu.
Time Frame: 21 days post-vaccination (Day 21)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influsplit SSW 2005/2006 10-13 Years Group
Number analyzed (Participants) | 75
Participants
  A/New Caledonia (H1N1), Dose 1: number analyzed (Participants) | 48
  A/New Caledonia (H1N1), Dose 1 | 33
  A/New York (H3N2), Dose 1: number analyzed (Participants) | 57
  A/New York (H3N2), Dose 1 | 52
  B/Jiangsu, Dose 1 | 62

8. Secondary Outcome: Number of Seroprotected Subjects Against 3 Strains of Influenza Disease in Children Aged Between 10 and 13 Years
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40. The three influenza strains assessed were: A/New Caledonia (H1N1), A/New York (H3N2), B/Jiangsu.
Time Frame: 21 days post-vaccination (Day 21)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influsplit SSW 2005/2006 10-13 Years Group
Number analyzed (Participants) | 106
Participants
  A/New Caledonia (H1N1), Dose 1 | 91
  A/New York (H3N2), Dose 1 | 101
  B/Jiangsu, Dose 1 | 93

9. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 4-day (Day 0-3) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects (with at least one vaccine administration documented) for whom data were available and who had a dairy card available. Post Dose 2 results are not available for the 10-13 years Group as these subjects received only one dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Influsplit SSW 2005/2006 6-9 Years Group | Influsplit SSW 2005/2006 10-13 Years Group
Number analyzed (Participants) | 110 | 114
Participants
  Pain, Any, Dose 1 | 62 | 54
  Pain, Grade 3, Dose 1 | 0 | 1
  Redness, Any, Dose 1 | 28 | 24
  Redness, > 50 mm, Dose 1 | 0 | 0
  Swelling, Any, Dose 1 | 28 | 39
  Swelling, > 50 mm, Dose 1 | 0 | 0
  Pain, Any, Dose 2: number analyzed (Participants) | 108 | 0
  Pain, Any, Dose 2 | 68 |
  Pain, Grade 3, Dose 2: number analyzed (Participants) | 108 | 0
  Pain, Grade 3, Dose 2 | 1 |
  Redness, Any, Dose 2: number analyzed (Participants) | 108 | 0
  Redness, Any, Dose 2 | 31 |
  Redness, > 50 mm, Dose 2: number analyzed (Participants) | 108 | 0
  Redness, > 50 mm, Dose 2 | 0 |
  Swelling, Any, Dose 2: number analyzed (Participants) | 108 | 0
  Swelling, Any, Dose 2 | 35 |
  Swelling, > 50 mm, Dose 2: number analyzed (Participants) | 108 | 0
  Swelling, > 50 mm, Dose 2 | 0 |
  Pain, Any, Across doses | 82 | 54
  Pain, Grade 3, Across doses | 1 | 1
  Redness, Any, Across doses | 39 | 24
  Redness, > 50 mm, Across doses | 0 | 0
  Swelling, Any, Across doses | 44 | 39
  Swelling, > 50 mm, Across doses | 0 | 0

10. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were Arthralgia, Fatigue, Fever, Headache, Myalgia, Shivering and Sweating. Any= occurrence of the symptom regardless of intensity grade. Grade 3 fever = Grade 3 symptoms greater than (>) 39.0 °C. Related = symptoms considered by the investigator to have a causal relationship to study vaccination.
Time Frame: During the 4-day (Day 0-3) post-vaccination period following each dose and across doses
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Influsplit SSW 2005/2006 6-9 Years Group | Influsplit SSW 2005/2006 10-13 Years Group
Number analyzed (Participants) | 110 | 114
Participants
  Arthralgia, Any, Dose 1 | 10 | 6
  Arthralgia, Grade 3, Dose 1 | 0 | 1
  Arthralgia, Related, Dose 1 | 9 | 6
  Fatigue, Any, Dose 1 | 22 | 22
  Fatigue, Grade 3, Dose 1 | 0 | 0
  Fatigue, Related, Dose 1 | 18 | 10
  Fever (Axillary), ≥ 37.5ºC, Dose 1 | 3 | 3
  Fever (Axillary), > 39.0ºC, Dose 1 | 0 | 0
  Fever (Axillary), Related, Dose 1 | 3 | 3
  Headache, Any, Dose 1 | 26 | 19
  Headache, Grade 3, Dose 1 | 0 | 1
  Headache, Related, Dose 1 | 19 | 10
  Myalgia, Any, Dose 1 | 22 | 13
  Myalgia, Grade 3, Dose 1 | 0 | 0
  Myalgia, Related, Dose 1 | 19 | 10
  Shivering, Any, Dose 1 | 10 | 8
  Shivering, Grade 3, Dose 1 | 0 | 1
  Shivering, Related, Dose 1 | 10 | 6
  Sweating, Any, Dose 1 | 2 | 4
  Sweating, Grade 3, Dose 1 | 0 | 0
  Sweating, Related, Dose 1 | 2 | 3
  Arthralgia, Any, Dose 2: number analyzed (Participants) | 108 | 0
  Arthralgia, Any, Dose 2 | 3 |
  Arthralgia, Grade 3, Dose 2: number analyzed (Participants) | 108 | 0
  Arthralgia, Grade 3, Dose 2 | 1 |
  Arthralgia, Related, Dose 2: number analyzed (Participants) | 108 | 0
  Arthralgia, Related, Dose 2 | 2 |
  Fatigue, Any, Dose 2: number analyzed (Participants) | 108 | 0
  Fatigue, Any, Dose 2 | 12 |
  Fatigue, Grade 3, Dose 2: number analyzed (Participants) | 108 | 0
  Fatigue, Grade 3, Dose 2 | 1 |
  Fatigue, Related, Dose 2: number analyzed (Participants) | 108 | 0
  Fatigue, Related, Dose 2 | 6 |
  Fever (Axillary), ≥ 37.5ºC, Dose 2: number analyzed (Participants) | 108 | 0
  Fever (Axillary), ≥ 37.5ºC, Dose 2 | 5 |
  Fever (Axillary), > 39.0ºC, Dose 2: number analyzed (Participants) | 108 | 0
  Fever (Axillary), > 39.0ºC, Dose 2 | 0 |
  Fever (Axillary), Related, Dose 2: number analyzed (Participants) | 108 | 0
  Fever (Axillary), Related, Dose 2 | 4 |
  Headache, Any, Dose 2: number analyzed (Participants) | 108 | 0
  Headache, Any, Dose 2 | 22 |
  Headache, Grade 3, Dose 2: number analyzed (Participants) | 108 | 0
  Headache, Grade 3, Dose 2 | 2 |
  Headache, Related, Dose 2: number analyzed (Participants) | 108 | 0
  Headache, Related, Dose 2 | 16 |
  Myalgia, Any, Dose 2: number analyzed (Participants) | 108 | 0
  Myalgia, Any, Dose 2 | 19 |
  Myalgia, Grade 3, Dose 2: number analyzed (Participants) | 108 | 0
  Myalgia, Grade 3, Dose 2 | 2 |
  Myalgia, Related, Dose 2: number analyzed (Participants) | 108 | 0
  Myalgia, Related, Dose 2 | 14 |
  Shivering, Any, Dose 2: number analyzed (Participants) | 108 | 0
  Shivering, Any, Dose 2 | 8 |
  Shivering, Grade 3, Dose 2: number analyzed (Participants) | 108 | 0
  Shivering, Grade 3, Dose 2 | 1 |
  Shivering, Related, Dose 2: number analyzed (Participants) | 108 | 0
  Shivering, Related, Dose 2 | 5 |
  Sweating, Any, Dose 2: number analyzed (Participants) | 108 | 0
  Sweating, Any, Dose 2 | 3 |
  Sweating, Grade 3, Dose 2: number analyzed (Participants) | 108 | 0
  Sweating, Grade 3, Dose 2 | 0 |
  Sweating, Related, Dose 2: number analyzed (Participants) | 108 | 0
  Sweating, Related, Dose 2 | 2 |
  Arthralgia, Any, Across doses | 13 | 6
  Arthralgia, Grade 3, Across doses | 1 | 1
  Arthralgia, Related, Across doses | 11 | 6
  Fatigue, Any, Across doses | 30 | 22
  Fatigue, Grade 3, Across doses | 1 | 0
  Fatigue, Related, Across doses | 22 | 10
  Fever (Axillary), ≥ 37.5ºC, Across doses | 7 | 3
  Fever (Axillary), > 39.0ºC, Across doses | 0 | 0
  Fever (Axillary), Related, Across doses | 6 | 3
  Headache, Any, Across doses | 38 | 19
  Headache, Grade 3, Across doses | 2 | 1
  Headache, Related, Across doses | 29 | 10
  Myalgia, Any, Across doses | 28 | 13
  Myalgia, Grade 3, Across doses | 2 | 0
  Myalgia, Related, Across doses | 23 | 10
  Shivering, Any, Across doses | 17 | 8
  Shivering, Grade 3, Across doses | 1 | 1
  Shivering, Related, Across doses | 14 | 6
  Sweating, Any, Across doses | 5 | 4
  Sweating, Grade 3, Across doses | 0 | 0
  Sweating, Related, Across doses | 4 | 3

11. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events.
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During 31 days after the study vaccine dose (Day 0-30)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects (with at least one vaccine administration documented) for whom data were available and who had a dairy card available.
Measure: Count of Participants; unit: Participants
Arm/Group | Influsplit SSW 2005/2006 6-9 Years Group | Influsplit SSW 2005/2006 10-13 Years Group
Number analyzed (Participants) | 110 | 114
Participants
  Subjects with any AE(s) | 52 | 30
  Subjects with Grade 3 AE(s) | 3 | 1
  Subjects with related AE(s) | 1 | 4

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period, from Day 0 to 58 + 5 days (30 + 5 days after the 2nd vaccine dose) for the 6-9 years Group and from Day 0 to 30 + 5 days (30 + 5 days after the vaccination) for the 10-13 years Group
Population: The analysis was performed on the Total Vaccinated Cohort, included all vaccinated subjects (with at least one vaccine administration documented) for whom data were available and who had a dairy card available.
Measure: Count of Participants; unit: Participants
Arm/Group | Influsplit SSW 2005/2006 6-9 Years Group | Influsplit SSW 2005/2006 10-13 Years Group
Number analyzed (Participants) | 110 | 114
Participants
  Any SAEs | 3 | 0
  Grade 3 | 0 | 0
  Related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general: during the 4-day (Day 0-3) post-vaccination period following each dose and across doses. Unsolicited adverse events (AEs): during 31 days after the study vaccine dose (Day 0-30). SAEs: during the entire study period, from Day 0 to 58 + 5 days (30 + 5 days after the 2nd vaccine dose) for the 6-9 years Group and from Day 0 to 30 + 5 days (30 + 5 days after the vaccination) for the 10-13 years Group.
Arm/Group | Influsplit SSW 2005/2006 6-9 Years Group | Influsplit SSW 2005/2006 10-13 Years Group
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/114
Serious Adverse Events (participants affected / at risk) | 3/110 | 0/114
Other Adverse Events (participants affected / at risk) | 100/110 | 90/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influsplit SSW 2005/2006 6-9 Years Group (N=110) | Influsplit SSW 2005/2006 10-13 Years Group (N=114)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hereditary fructose intolerance (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influsplit SSW 2005/2006 6-9 Years Group (N=110) | Influsplit SSW 2005/2006 10-13 Years Group (N=114)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (3)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 6 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Chills (General disorders) | 17 (18) | 8 (8)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 4 (5) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 39 (59) | 24 (24)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 30 (34) | 22 (22)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (2) | 2 (2)
Headache (Nervous system disorders) | 38 (50) | 19 (20)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1)
Lice infestation (Infections and infestations) | 2 (2) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (41) | 13 (13)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Otosalpingitis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 82 (130) | 54 (54)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 11 (12) | 4 (4)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 7 (8) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 3 (3) | 0 (0)
Swelling (General disorders) | 44 (63) | 39 (39)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 13 (14) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.